CLINICAL TRIAL: NCT04168242
Title: The Psychological Impact of Scalp Cooling in Patients Receiving Chemotherapy for Primary Gynecologic Cancers: a Randomised Trial
Brief Title: Scalp Cooling in Gynecologic Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UWB 19-514
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-10

CONDITIONS: Gynecologic Cancer; Chemotherapy-Induced Change
Keywords: Gynecologic cancer; chemotherapy-induced alopecia; scalp cooling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Patients have scalp cooling during the chemotherapy period
  Interventions: Device: Scalp cooling Paxman Orbis II system
- Control arm (Placebo Comparator): Patients do not have scalp cooling during the chemotherapy period
  Interventions: Other: Standard treatment

INTERVENTIONS:
Device: Scalp cooling Paxman Orbis II system — The experimental arm will have scalp cooling that starts 30 minutes before the chemotherapy, continues throughout the infusion of the chemotherapy, and lasts for 20-90 minutes more depending on the type of regimen.
  Arms: Experimental arm
Other: Standard treatment — The control arm will not have scalp cooling before, during and after chemotherapy.
  Arms: Control arm

SUMMARY:
In gynecologic cancers, many common chemotherapy agents can lead to chemotherapy-induced alopecia. Currently scalp cooling is the most well studied preventive measure. However, its acceptability and its impact on patients' QOL in Asian population is unclear.

DETAILED DESCRIPTION:
Dynamic scalp cooling system prevents alopecia by inducing vasoconstriction leading to a reduction of scalp blood flow, thus reducing the delivery of cytotoxic drugs to the hair follicles and reducing follicular metabolic activities. One recent meta-analysis included 10 studies showed that the efficacy was 43% in general.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years old.
2. Patients with primary gynecologic cancers.
3. Patients who are going to receive at least four cycles of chemotherapy that are known to induce alopecia, such as carboplatin, paclitaxel, taxotere, topotecan, etoposide, vincristine and ifosfamide.
4. Patients who are fit to give informed consent.

Exclusion Criteria:

1. Patients who have pre-existing alopecia of CTCAE v5.0 grade 1 or above will be excluded.
2. Patients who have the following conditions will be excluded:

   1. migraine
   2. scalp or brain metastasis
   3. hypothyroidism
   4. uncontrolled diabetes
   5. liver and / or renal derangement (where liver enzymes and / or creatinine are 1.5x more than upper normal limit)
   6. severe untreated anaemia
   7. cold sensitivity
   8. cold agglutinin disease, cryoglobulinemia, or cryofibrinogenemia
3. Patients who had brain irradiation.
4. Patients who have documented psychiatric disorders will be excluded.
5. Patients who are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence and grading of chemotherapy induced alopecia | 9 months
  Will be assessed by Dean's scale Grade 0 - 4 (from 0% to >75% hair loss)

SECONDARY OUTCOMES:
Quality-of-life scale | 9 months
  Different functional scales will be assessed by questionnaires like the EORTC questionnaires where all scales range from 0-100. The higher the score, the greater the intensity of that particular item is.
Anxiety / depression level | 9 months
  Anxiety and depression scales will be assessed by GAD7 PHQ9. A higher score means the more frequent an event is.
Incidence and grading of treatment-related adverse events | 9 months
  Will be assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yu Tse, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong